CLINICAL TRIAL: NCT05086315
Title: An Open-label, First-in-human, Dose-escalation/Expansion Study of SAR443579 Administered as Single Agent by Intravenous Infusion in Adult and Pediatric Participants With Relapsed or Refractory Acute Myeloid Leukemia (R/R AML), B-cell Acute Lymphoblastic Leukemia (B-ALL), High Risk-myelodysplasia (HR-MDS), or Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Brief Title: First-in-human Study of SAR443579 Infusion in Male and Female Children and Adult Participants With Relapsed or Refractory Acute Myeloid Leukemia (R/R AML), B-cell Acute Lymphoblastic Leukemia (B-ALL), High Risk-myelodysplasia (HR-MDS), or Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD17197; U1111-1266-7399 (Registry Identifier: ICTRP); 2023-508357-58 (Registry Identifier: CTIS); 2021-004287-98 (EudraCT Number)
Record Dates: First submitted 2021-10-19; First posted 2021-10-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphocytic Leukaemia; Acute Myeloid Leukaemia Refractory; Myelodysplastic Syndromes; Blastic Plasmacytoid Dendritic Cell Neoplasia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR443579 (Experimental): Dose Escalation: SAR443579 administered intravenously at escalating dose levels.
  Dose Expansion: SAR443579 administered intravenously at the recommended dose and schedule determined from the dose escalation.
  Interventions: Drug: SAR443579

INTERVENTIONS:
Drug: SAR443579 — Powder for solution for infusion; by IV infusion

SUMMARY:
This is an open-label, multicenter, Phase 1/Phase 2, dose escalation and dose expansion study to evaluate the safety, pharmacokinetics, pharmacodynamics and anti-leukemic activity of SAR443579 in various hematological malignancies.

DETAILED DESCRIPTION:
Study duration per participant is 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 1 year (for France: 2 years) old at the time the trial participant or legal guardian signs the informed consent form and will be assigned as follows:

  * Adult arm: aged at least 18 years old.
  * Pediatric arm: aged 1 (for France: 2 years) to less than 18 years old.
* Adult and Pediatric Arms: Escalation and Expansion/Optimization Cohorts A1, A2, C, D: Confirmed diagnosis of primary or secondary AML (any subtype) according to World Health Organization (WHO) 2022 classification. Participants with AML must meet one of the following criteria, a), b), c) or d) and are limited to those with no available (or are ineligible) therapy with known clinical benefit.

  a) Primary Induction Failure (PIF) AML, defined as disease refractory to one of the following, i or ii.

  i) An intensive induction attempt, per institution. Induction attempts include high-dose and/or standard-dose cytarabine ± an anthracyclines/anthracenedione ± an anti-metabolite, with or without growth factor or targeted therapy containing regimens.

ii) For adults who are age 75 years or older, or who have comorbidities that preclude use of intensive induction chemotherapy; PIF is defined as AML refractory to one of the following less intensive regimens, 1 or 2:

1. 4 cycles of hypomethylating agents (HMA) or
2. 2 cycles HMA + venetoclax b) Early relapse (ER) AML, defined as AML in relapse with CR, CRh or CRi duration less than 6 months on prior induction treatment c) Leukemia in first or higher relapse d) For participants aged 1 (for France: 2 years) to less than 18 years old, primary induction failure is defined as disease refractory after two cycles of induction therapy.

   * Adult Arm (Escalation and Expansion/Optimization Cohorts B and Japan Cohort C only): Confirmed diagnosis of MDS, meeting the following criteria:

     1. intermediate or high-risk category as per a Revised International Prognostic Scoring System (IPSS-R) AND
     2. confirmed CD123 + expression status determined by local institutional standards AND
     3. limited to those with no available (or are ineligible) therapy with known clinical benefit.
   * Pediatric arms escalation part and Japan Cohort C only: Confirmed diagnosis of CD123+ BALL without extramedullary lesions that have no available (or are ineligible) therapy with known clinical benefit. Participants with non-CNS chloromatous disease are not allowed in the study.
   * Body weight at least 10 kg.
   * Pediatric arm and escalation part only: Confirmed diagnosis of BPDCN according to World Health Organization (WHO) 2022 classification, who have relapsed or refractory disease with no available (or are ineligible) therapy with known clinical benefit.
   * Japan participants (Cohort C): Participant must be at least 18 years old at the time the trial participant signs the informed consent form

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status greater than 2 (at least 18 years-old). Karnofsky Scale (16 to 17 years-old) less than 50% or Lansky Scale (less than 16 years-old) less than 50%.
* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that requires or required treatment with systemic immunosuppressive treatments, which may suggest a risk for immune-related adverse events. The following are not exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that required only hormone replacement or psoriasis that does not require systemic treatment.
* History of an invasive malignancy within the last 3 years prior to first IMP administration that requires active therapy (adjuvant hormonal therapy is allowed) other than the one treated in this study.
* Evidence of active central nervous system leukemia at the time of enrollment as evidenced by cytology or pathology. Except for participants aged 1 (for France: 2 years) to less than 18 years, central nervous system 1 disease (CNS1) and CNS2 disease are allowed.
* Known acquired immunodeficiency syndrome (AIDS-related illnesses) or human immunodeficiency virus (HIV) disease requiring antiretroviral treatment, or having active hepatitis B or C infection, or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Prior treatment with an anti-CD123-directed agent (except for participants with BPDCN in the pediatric arm).
* Prior HSCT with relapse beyond 3 months or prior CAR-T therapy in B-ALL with relapse beyond 2 months may be included only if off immunosuppression for a minimum of 4 weeks and no evidence of GVHD.
* Receiving at the time of first investigational medicinal product (IMP) administration corticosteroid as a concomitant medication with corticosteroid dose more than 10 mg/day of oral prednisone or the equivalent.
* AML, BPDCN, or HR-MDS participants with prior treatment with cellular therapy, eg, chimeric antigen receptor T cell (CAR-T) or chimeric antigen receptor NK cell (CAR-NK). Prior CAR-T therapy is allowed for participants with B-ALL.
* Concurrent treatment with other investigational drugs.
* Pregnant and breast-feeding women.
* History of solid organ transplant, including corneal transplant.
* Average QTc (using the Fridericia correction calculation) greater than 470 millisecond (msec) at screening.
* Pediatric arm only: Participants with known inherited bone marrow failure syndromes (e.g., bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome). Participants with Down syndrome with adequate organ function as per Investigator discretion are allowed to participate in the study.
* Adult arm Expansion/Optimization- Participants with MDS evolving from a pre-existing myeloproliferative neoplasm (MPN), MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), unclassifiable MDS/MPN and therapy-related MDS (t-MDS).
* Confirmed diagnosis of acute promyelocytic leukemia (APL) or juvenile myelomonocytic leukemia (JMML) according to WHO 2022 classification.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Escalation Part: Incidence of dose-limiting toxicity (DLT) | Day 1 to Day 28
  DLTs encompass both hematologic and nonhematologic toxicities, prespecified adverse reactions observed post-administration of SAR443579 and assessed by both the investigator and the sponsor.
Japan Cohort C: Incidence of DLT in Japanese participants | Day 1 to Day 28
  DLTs encompass both hematologic and nonhematologic toxicities, prespecified adverse reactions observed post-administration of SAR443579 and assessed by both the investigator and the sponsor.
Expansion/Optimization part (Cohorts A1, A2 & D), AML: Proportion of participants who have a CR + CRh + CRi according to the modified AML IWG 2003 criteria | Up to 6 months
  Measure of clinical response to treatment: Proportion of participants who have a complete remission (CR) + CR with partial hematologic recovery (CRh) + CR with incomplete hematologic recovery (CRi) according to the modified acute myeloid leukemia (AML) IWG 2003 criteria.
Expansion/Optimization part (Cohort B), MDS: Overall response rate (CR + CR equivalent + PR + CRL + CRh + HI) according to the IWG 2023 MDS response criteria | Up to 6 months
  Measure of clinical response to treatment: Overall response rate (CR + CR equivalent + partial remission (PR) + CR with limited count recovery (CRL) + CRh + hematologic improvement (HI)) according to the International Working Group (IWG) 2023 myelodysplasia (MDS) response criteria.

SECONDARY OUTCOMES:
Expansion/Optimization part - Cohorts A, B and D: Recommended dose for expansion (RDE) | Up to 12 months
  Recommended dose for expansion (RDE) of SAR443579.
Escalation and Expansion/Optimization parts - Cohorts A, B, C and D: Number of participants with TEAEs | Up to 30 months
  Number of participants with treatment-emergent adverse events (TEAEs).
Cohorts A, B, C and D: Ctrough at Cycle 1 | Cycle 1 from Day 1 to Day 28
  Concentration observed just before treatment administration during repeated dosing (Ctrough).
Cohorts A, B, C and D: Incidence of ADA | Up to 30 months
  Percentage of participants with anti-drug antibody (ADA) against SAR443579.
Escalation and Expansion/Optimization parts - Japan Cohort C, AML: Rate of CR + CRh + CRi per AML 2003 modified IWG response criteria | Up to 6 months
  Measure of clinical response to treatment.
Escalation and expansion/Optimization parts - Japan Cohort C, MDS: CR rate and ORR rate per IWG 2023 MDS response criteria for escalation part and ORR rate per IWG 2023 | Up to 6 months
  Measure of clinical response to treatment.
Escalation and Expansion/Optimization parts - Japan Cohort C, B-ALL: Rate of CR + CRh + CRi as defined by National Comprehensive Cancer Network (NCCN) | Up to 6 months
  Measure of clinical response to treatment.
Expansion/Optimization part - Cohorts A and D: Overall response rate (ORR) | Up to 6 months
  Measure of clinical response to treatment.
Expansion/Optimization part - Cohorts A and D: Duration of CR + CRh + CRi (Duration of CRc) | Up to 30 months
  Measure the length of clinical response to treatment.
Expansion/Optimization part - Cohorts A and D: Duration of CR + CRi + CRh + PR + MLFS (Duration of overall response rate) | Up to 30 months
  Measure the length of clinical response to treatment.
Expansion/Optimization part - Cohorts A and D: Alternative CR rate | Up to 6 months
  Measure of clinical response to treatment.
Expansion/Optimization part - Cohorts A and D: Duration of CR + CRh (Duration of alternative CR) | Up to 30 months
  Measure the length of clinical response to treatment.
Expansion/Optimization part - Cohorts A and D: Event-free survival (EFS) | Up to 6 months
  EFS is defined as the time interval from the first day of treatment assignment to the date of earliest evidence of relapse, treatment failure, or death.
Expansion/Optimization part - Cohorts A and D: Overall survival (OS) | Up to 30 months
  OS is defined as time interval from the first day of treatment assignment to death from any cause.
Expansion/Optimization part - Cohorts A and D: Rate of hematopoietic stem cell transplantation (HSCT) | Up to 30 months
  Rate of HSCT procedures immediately following study treatment administration but prior to subsequent therapy for treatment of AML.
Expansion/Optimization part - Cohorts A and D: Time to treatment failure (TTF) | Up to 6 months
  TTF is defined as the time from first day of treatment assignment to discontinuation for any reason excluding remission, eg, relapsed disease, refractory disease, unacceptable AE, participant preference or death.
Expansion/Optimization part - Cohorts A and D: Rate of conversion from transfusion dependence | Day 0 to Day 56
  Rate of conversion from transfusion dependence during 56-day post-baseline period.
Expansion/Optimization part - Cohorts A and D: Rate of participants who are transfusion independent at baseline and remain independent during 56-day postbaseline period | Day 0 to Day 56
  Rate of participants who are transfusion independent at baseline and remain independent during 56-day postbaseline period.
Expansion/Optimization part - Cohort B: Alternative CR rate | Up to 6 months
  Alternative CR rate defined as proportion of participants with CR, CR equivalent, CRuni, CRbi, and CRh.
Expansion/Optimization part - Cohort B: Duration of ORR | Up to 30 months
  The time interval from the first documented evidence of CR, CR equivalent, CRL, CRh, PR or HI to PD or relapse from CR, CR equivalent, CRL, CRh, PR or HI as per 2023 IWG recommendations or death due to any cause, whichever comes first.
Expansion/Optimization part - Cohort B: Event-free survival (EFS) | Up to 30 months
  EFS is defined as the time interval from the first day of treatment assignment to the date of protocol specified events.
Expansion/Optimization part - Cohort B: Overall survival (OS) | Up to 30 months
  OS is defined as time interval from the first day of treatment assignment to death from any cause.
Expansion/Optimization part - Cohort B: Rate of hematopoietic stem cell transplantation (HSCT) | Up to 30 months
  Rate of HSCT procedures immediately following study treatment administration but prior to subsequent therapy.
Expansion/Optimization part - Cohort B: Time to treatment failure (TTF) | Up to 30 months
  TTF is defined as the time interval from first day of treatment assignment to discontinuation for any reason excluding remission, eg, relapsed disease, disease progression, unacceptable AE, participant preference or death.
Expansion/Optimization part - Cohort B: Duration of alternative CR (CR + CR equivalent + CRL + CRh) | Up to 30 months
  Measure the length of clinical response to treatment.
Expansion/Optimization part - Cohort B: Progression free survival (PFS) | Up to 30 months
  The time interval from the first day of treatment assignment to the date of PD, relapse from CR (or CR equivalent), PR, CRL, CRh, or HI, death due to any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- United States (10):
  - City of Hope-Site Number:8400002, Duarte, California
  - Emory University School of Medicine- Grady Campus- Site Number : 8400006, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center-Site Number:8400004, Boston, Massachusetts
  - Weill Cornell Medical College-Site Number:8400003, New York, New York
  - Montefiore Hutchinson Campus- Site Number : 8400012, The Bronx, New York
  - The Ohio State University- Site Number : 8400009, Columbus, Ohio
  - Oregon Health and Science University-Site Number:8400011, Portland, Oregon
  - The Children's Hospital of Philadelphia- Site Number : 8400013, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center-Site Number:8400001, Houston, Texas
  - Seattle Children's Hospital- Site Number : 8400014, Seattle, Washington
- Australia (2):
  - Investigational Site Number :0360002, Melbourne, Victoria
  - Investigational Site Number :0360001, Melbourne, Victoria
- China (2):
  - Investigational Site Number : 1560001, Tianjin
  - Investigational Site Number : 1560003, Zhengzhou
- France (4):
  - Investigational Site Number :2500002, Marseille
  - Investigational Site Number :2500001, Paris
  - Investigational Site Number : 2500004, Paris
  - Investigational Site Number :2500003, Villejuif
- Netherlands (5):
  - Investigational Site Number :5280002, Amsterdam
  - Investigational Site Number :5280003, Groningen
  - Investigational Site Number : 5280005, Nijmegen
  - Investigational Site Number :5280001, Rotterdam
  - Investigational Site Number :5280004, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TCD17197 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25348&tenant=MT_SNY_9011